CLINICAL TRIAL: NCT06170073
Title: Hong Kong Cohort of Abnormal Sleep in Ageing Population (HK-ASAP): an Observational Study on Brain Health and Sleep Quality in Community-dwelling Older Adults
Brief Title: Hong Kong Cohort of Abnormal Sleep in Ageing Population (HK-ASAP): Focusing on Brain Health and Sleep Quality
Acronym: HK-ASAP
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2023.496
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sleep Disturbance; Aging; Cognitive Decline; Brain Disease
Keywords: Ageing; Sleep disturbances; Cognition; Brain health; Longevity
MeSH Terms: conditions — Parasomnias; Cognitive Dysfunction; Brain Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participant's saliva will be collected for further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Poor sleepers: With a total score of Pittsburgh Sleep Quality Index (PSQI) > 5.
- Good sleepers: With a total score of Pittsburgh Sleep Quality Index (PSQI) ≤ 5.

SUMMARY:
Poor sleep quality can significantly jeopardize the brain health, cognitive functions, daily activities, quality of life, and even be implicated as a key potential contributing factor in the development of accelerated cognitive decline and prodromal dementia. Consequently, research efforts to understand, and therefore potentially model, the effects of sleep quality on cognition and brain health are of great pragmatic values.

DETAILED DESCRIPTION:
Objectives: This study aims to investigate the cognitive changes in older adults with sleep disturbances, examine the neuroimaging contributors to poor sleep quality and cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

* Chinese old adults are the ones who are over 60 years of chronological age.
* Sleep disturbance: individual's subjective sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI) with a total score >5.

Exclusion Criteria:

* History of bipolar disorders or psychosis.
* History of major neurological deﬁcits, including stroke, transient ischemic attack or brain tumor.
* Unable to participant magnetic resonance imaging (MRI) scanning.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normal ageing adults and adults with sleep disturbances.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Pittsburgh Sleep Quality Index (PSQI) is a validated 19-item self-reported questionnaire
Global cognition will be measured by the Montreal Cognitive Assessment Hong Kong version (HK MoCA) | Baseline
  The Montreal Cognitive Assessment Hong Kong version (HK MoCA) is a validated and widely used screening assessment for detecting cognitive impairment, which measures an array of cognitive functions such as visuospatial, memory, language and attention.
Complex attention will be measured by the Attention Network Test (ANT) | Baseline
  The ANT paradigm, as a computerized test, was used and performed by E-Prime 3.0.

SECONDARY OUTCOMES:
Memory and learning will be measured by the Word list learning test (WLLT) | Baseline
  Word list learning test (WLLT), consisting of fifteen semantically non-associated words that is presented consecutively over three free trials of immediate recall, a 20-min delayed recall and followed by yes/no recognition.
Executive functions will be measured by the category verbal fluency test (CVFT) | Baseline
  On each trial of CVFT, the participants will be asked to overtly generate words in the animal category, fruit category and vegetable category as many as possible within 60 seconds
The levels of Aβ40 and Aβ42 will be measured by saliva analysis | Baseline
  saliva samples will be collected at a consistent time of day to avoid circadian effects and will be kept on ice during the collection.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna LU, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Tai Po District, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided